CLINICAL TRIAL: NCT00688220
Title: Effect of Celliant Materials on Pain and Blood Oxygenation in Subjects With Chronic Elbow and Wrist Pain
Status: Terminated | Type: Observational
Why Stopped: PI closed study due to lack of enrollment
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Hologenix, LLC (Industry)
Responsible Party: Ian Gordon, M.D., Ph.D., VA Long Beach Healthcare System
Other Study IDs: #887
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Wrist Pain; Chronic Elbow Pain
Keywords: Arthritis; Carpel tunnel syndrome; Epicondylitis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Those wearing garments fabricated with Celliant
- 2: Those not wearing garments fabricated using Celliant (placebo).

SUMMARY:
The purpose of this research is to determine whether a new type of fabric, Celliant, can reduce elbow and wrist pain associated with chronic medical conditions such as carpel tunnel syndrome, arthritis or tennis elbow and whether it can increase blood flow and oxygenation levels in the arms and hands after wearing the material.

DETAILED DESCRIPTION:
A new type of fabric, Celliant, is made from polymer yarns containing optically active particles (1-1.2 micron diameter titanium dioxide, quarts and aluminum oxide particles) with modify absorption, reflection and transmission of light in the visible and near infrared portion of the spectrum. It is believed that the Celliant particles increase skin illumination such taht cytochrome pigments and other enzymes are activated, leading to increased blood flow and oxygenation of the skin and neighboring soft tissues. In addition, numerous anecdotal reports from patients with chronic foot and arm pain indicate that wearing Celliant garments for even a few days leads to dramatic improvement in many different painful conditions. This is a single center, stratified, randomized, prospective, double-blind study. Questionnaires that subjects will be asked complete are 1) Visual Analog Scale, 2) Brief Pain Inventory, 3) McGill Short Form Pain Survey and 4) SF-36 Quality of Life Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain for a minimum of 6 months
* A score of equal to or greater than 3 on question III of McGill Short Form Pain Questionnaire

Exclusion Criteria:

* Open wounds on the involved limb
* Threatened limb loss from ischemia
* Changes in pain or inflammatory medication within the last 30 days
* Psychiatric or other conditions that would affect compliance
* Inability to comply with use of the study articles or to fill out questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating subjects will be recruited who have chronic elbow or wrist pain from epidondylitis, carpal tunnel syndrom or other chronic disease - 40 with chronic elbow and 40 will chronic wrist pain.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mean questionnaire scores for each question at Visits 1 and 2 will be compared to the mean scores from Visits 3 and 4 to assess change in symptoms in subjects with Celliant or placebo garments using Mann-Whitney t-test statistics. | 4 weeks
Oxygenation levels of the elbow or wrist and hands at each time point will be compared between Celliant and placebo materials using standard statistical methods | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gordon, M.D., Ph.D., Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States